CLINICAL TRIAL: NCT02263560
Title: Supraspinal Contributions to the Control of Human Locomotion: Clinical and Fundamental Aspects
Acronym: SUPLOCO
Status: Completed | Type: Observational
Sponsor: University of Fribourg (Other)
Collaborators: Dr Titus Bihl, Hopital Cantonal Fribourgeois (Unknown)
Responsible Party: Principal Investigator, Halim HICHEUR, Lecturer (PhD), University of Fribourg
Other Study IDs: UFribourg
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Post-stroke Gait Assessments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (2):
- Post-stroke patients: Patients who experienced stroke and who already recover gait abilities.
  Interventions: Behavioral: Kinematic measurements
- Control population: Participants matching the criterion (age and gender) of the patients' group.
  Interventions: Behavioral: Kinematic measurements

INTERVENTIONS:
Behavioral: Kinematic measurements

SUMMARY:
Many neurological patients express enhanced deficits while walking in a dark room (or during the night): the supraspinal structures involved in this navigational deficit have not been identified yet. In this project, the investigators will study post-stroke gaits of human patients and compare them to those of a control population during a goal-oriented task performed in different visual conditions.

The investigators want to test the hypothesis that during simple goal-oriented locomotor tasks, only patients with specific (e.g. medio or infero- temporal) lesions will express navigational deficits.

ELIGIBILITY:
Inclusion Criteria (for matching controls):

* Adult male and female subjects (18-->85 years old)

Exclusion Criteria (for matching controls):

* Persons with history of an acquired or congenital neurological disorder, e.g. stroke, multiple sclerosis, Parkinson disease, increased intracranial pressure, etc.;
* Persons injured at the time of the experiments (fractures,…);
* Persons having reported repetitive spatial troubles/disorders;
* Persons with eye disorders and non-corrected vision problems;
* Pregnant women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The selected patients will be described by following parameters:
  * Parameters in relation to the person: age, gender.
  * Parameters in relation to the pathology: NIHSS, exact localisation, time since start of the symptoms, FIM (functional independence measure) visual field (ophthalmological examen), visual acuity (ophtalmological examen), visual neglect (Bells Cancellation Task), visuo-spatial short term working memory (Corsi span), visual motor integration (3-D cub subtest MoCA)
  * Parameters in relation to hospital stay: length of stay.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Walking stability indices of post-stroke patients | 1 hour and 30 minutes (including pre-tests, instructions delivery...).
Spatial accuracy of walking trajectories in post-stroke patients | 1 hour and 30 minutes (including pre-tests, instructions delivery...).

CONTACTS AND LOCATIONS:
Locations (1):
- University (UNIFR) and Hospital of Fribourg (HFR), Fribourg, Switzerland